CLINICAL TRIAL: NCT06101745
Title: Phase 2/3 Randomized Controlled Semi-blinded Trial to Investigate Safety and Effectiveness in Ureter Visualization With Intravenous Nizaracianine Triflutate, in up to 3 Divided Doses, in Adults Undergoing Abdominopelvic Surgery (TRIPHASE)
Brief Title: Trial to Visualize the Ureters With Nizaracianine Triflutate in Adults Undergoing Abdominopelvic Surgery
Acronym: TRIPHASE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Curadel Surgical Innovations, Inc. (Industry)
Collaborators: Leiden University Medical Center (Other); Erasmus Medical Center (Other); University of Massachusetts Chan Medical School, Worcester (Unknown); Stanford University (Other); Cedars-Sinai Medical Center (Other); University Medical Center Groningen (Other); Martini Hospital Groningen (Other); Isala (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ZW800-001
Record Dates: First submitted 2023-10-13; First posted 2023-10-26 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Injury of Ureter During Surgery (Disorder)
Keywords: Nizaracianine Triflutate; ZW800-1; ureter; ureter visualization; abdominopelvic surgery; Near-infrared; fluorescence imaging; TRIPHASE
MeSH Terms: interventions — ZW800-1 compound; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nizaracianine Triflutate Study Drug Arm (Active Comparator): Participants will receive up to 3 intravenous bolus injections with a minimal interval between doses of 60 minutes (surgeon discretion). Dose will be 1.0 or 2.5 mg depending on trial phase.
  Interventions: Drug: Nizaracianine Triflutate
- Sugar Comparator Arm (Placebo Comparator): In Phase 3A only, ~50 subjects will be randomly allocated to receive sugar placebo.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Nizaracianine Triflutate — Participants will receive up to 3 intravenous bolus injections with a minimal interval between doses of 60 minutes (surgeon discretion). Dose will be 1.0 or 2.5 mg depending on trial phase.
  Other Names: ZW800-1
  Arms: Nizaracianine Triflutate Study Drug Arm
Drug: Placebo Comparator — In Phase 3A only, ~50 subjects will be randomly allocated to receive sugar placebo
  Other Names: Sugar
  Arms: Sugar Comparator Arm

SUMMARY:
The goal of this clinical trial is to determine if the drug Nizaracianine Triflutate can help surgeons see and avoid the ureters during abdominopelvic surgery. The ureters are thin-wall, collapsible tubes that connect the kidneys to the bladder. They are difficult to see during surgery and are sometimes damaged accidentally. The main questions to answer are: 1) is this drug safe for use in patients undergoing abdominopelvic surgery and 2) can the drug see the ureters while simultaneously providing information about how well they are working. The clinical trial has 3 parts. Surgery patients enrolled in the first part (Phase 2) will receive drug at different doses to determine the best dose. Patients enrolled in the second part (Phase 3A) will be randomly assigned to drug or placebo (sugar), at the best dose from Phase 2, so the two can be compared directly. Patients enrolled in the final part (Phase 3B) will all receive drug at the best dose from Phase 2.

DETAILED DESCRIPTION:
Human surgery often suffers from poor visual contrast among anatomical landmarks within the surgical field and distinguishing one anatomical structure from another becomes nearly impossible if covered by connective tissue, blood, and/or bodily fluids.

A major unsolved problem in surgical imaging is anatomical enhancement of the ureters. Damage to the ureters is a serious unintended complication of abdominopelvic and retroperitoneal surgery, with rates as high as 30% in certain gynecological procedures. Ureter damage also leads to extraordinarily high patient morbidity and cost. Currently, to avoid this complication during certain surgeries involving the ureters, much time is taken to define their anatomy using meticulous tissue dissection. Even with such special care, though, approximately 80% of ureteral injuries are only discovered post-operatively when dramatic clinical signs emerge such as rigor, fever, abdominal pain, and/or bacteremia.

Ureter injury disproportionally impacts women, not only because of gynecological procedures but some reports have indicated female gender appears to predispose to injury during colectomies. Thus, the lack of availability of a safe diagnostic agent to provide real-time identification of the ureters and assessment of ureter function contributes to the gender disparity that exists within healthcare. Furthermore, patients in non-urban settings may not have access to surgeons with a large surgical volume and thus the years of specialized experience necessary to avoid ureter damage. Surgeon inexperience was identified as a prime risk factor for ureter injury, and teaching hospitals have been implicated in having an increased risk for ureter injury as well.

Visual contrast enhancement of the ureters should provide enormous benefit to both patient and surgeon including more rapid initial identification, continuous real-time mapping, reducing or elimination the need for surgical dissection and associated complications in some cases, reducing anesthesia time, and reducing the risk of iatrogenic damage during abdominopelvic procedures across all patient populations. And, if iatrogenic damage still occurs, visual contrast enhancement can quickly identify the site of injury so appropriate repair can be initiated intraoperatively.

Nizaracianine Triflutate (ZW800-1) is a novel small molecule drug with a unique zwitterionic chemical structure. This structure prevents the drug from binding non-specifically to tissues and organs after injection and facilitates its excretion by the kidneys into urine. Once in urine, Nizaracianine Triflutate creates visual contrast in the ureters that would otherwise not exist, and using a near-infrared (NIR) camera, surgeons can find the ureters and assess their function in real-time.

The clinical trial is divided into three parts:

Phase 2 originally planned to test 3 different doses of Nizaracianine Triflutate in 12 subjects per dose. The planned Phase 2 cohort 3 (5 mg per dose x3 for a total of 15 mg) was removed in the current version of the protocol as available results from the 1 mg cohort and 2.5 mg cohort indicated that the ureters could be readily visualized and there was an anticipated high risk of NIR camera saturation with the 5 mg dose. The Lead PI determined that there was no scientific or clinical justification to escalate to a 5 mg dose in the Phase 2 portion of the study. Each of the subjects in the other 2 cohorts received a total of 3 injections of the drug during surgery so that the ureters were visualized throughout. At the end of Phase 2, the best dose for imaging the ureters was selected as 2.5mg Nizaracianine Trifluatate.

Phase 3A will use 2.5mg Nizaracianine Trifluatate and will randomize ~100 subjects total, stratified for re-operative/inflammatory bowel status and BMI, then randomized 1:1 to treatment and control arms, to receive either placebo (sugar) or Nizaracianine Triflutate. Surgeon and subject will be blinded to what is administered.

Phase 3B will also use 2.5mg Nizaracianine Trifluatate and will administer drug to ~200 subjects. All subjects will receive the drug and surgeons can administer it up to three times depending on the length of the surgery, with each subject serving as their own control by comparing white light to NIR light.

During all three parts of the trial, safety of the drug will be monitored closely.

The long-term goal of this Phase 2/Phase 3 clinical trial is to determine whether Nizaracianine Triflutate provides the surgeon with visualization of the ureters throughout surgery, and in so doing can help them lower the risk of injury and improve patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Scheduled to undergo a medically necessary abdominopelvic surgical procedure expected to last ≥ 2 hours (Phase 2) or any duration (Phase 3), during which one or more ureters should be visualized during the procedure. All abdominopelvic surgical procedures are eligible unless specifically excluded in the Exclusion Criteria.
* For Phase 2, the procedure must require identification of one or both ureters using dissection, mobilization, or other surgical means.
* The planned surgical procedure is open or minimally invasive surgery (MIS), including robotic.
* Both ureters are expected to be present and functional.
* Capable and willing to provide informed consent prior to study-specific procedures
* Screening laboratory test results are within normal limits, or if any are outside of normal limits, they are considered by the site PI, and confirmed by the lead PI, to be clinically insignificant.
* Negative pregnancy test in women of childbearing potential

Exclusion Criteria:

* Known cardiovascular or pulmonary disease, renal or liver dysfunction, immunological disease, diabetes, or active cancer that would render the study subject unfit for surgery
* The planned surgical procedure is renal transplant or nephrectomy [note: partial nephrectomy is permitted provided that estimated glomerular filtration rate (eGFR) is not expected to fall below normal age-based limits]
* Prior renal transplant
* Impaired renal function defined as an estimated glomerular filtration rate (eGFR) < 50 mL/min/1.73m2
* Impaired liver function defined as values > 1.5 times the upper limit of normal (ULN) for alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), and total bilirubin, or < lower limit of normal (LLN) for albumin
* Coagulopathy as manifested by international normalized ration (INR) > 1.3 (unless patient is on anti-coagulants)
* Subjects with a marked baseline prolongation of QT/ corrected QT interval (QTc) interval (e.g., a QTc interval > 480 msec [CTCAE grade 1] using Fridericia's QT correction factor (14)
* History of a clinically significant allergy or anaphylaxis to a component of the investigational medicinal product (IMP)
* Known sensitivity to fluorescent light
* Alcohol or recreational drug use that meets diagnostic and statistical manual of mental disorders (DSM5) criteria for moderate or severe substance use disorder
* Pregnant or breastfeeding, or lack of effective contraception for at least one week post-surgery in male or female subjects with reproductive potential: for males, condom use; for females, oral contraceptives, diaphragm, or intrauterine devices (IUDs)
* Any condition that the investigator considers to be potentially jeopardizing to the study subject's well-being or the study's objectives.
* Participated in an interventional clinical research study within the previous 30 days.
* The planned use of an 800 nm NIR fluorophore that is not Nizaracianine (e.g., indocyanine green or Pafolacianine) immediately before, during, or immediately after the planned abdominopelvic procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The fraction of subjects for whom the surgeon is able to successfully identify the required length of the ureters (specified by the surgeon at each timepoint), as verified by three independent blinded reviewers. | 1 day (day of surgery)
  The proportion of subjects for whom the surgeon is able to successfully identify the required length of the ureters (specified by the surgeon at each timepoint) with a peak signal-to-background ratio (SBR) ≥ 1.5 where SBR is signal-to-background ratio - verified by three independent blinded reviewers

SECONDARY OUTCOMES:
The fraction of cases in which ureter identification did not require invasive procedures or dissection of surrounding tissue | 1 day (day of surgery)
  Measure the fraction of cases in which ureter identification did not require invasive procedures or dissection of surrounding tissue
Average time required for initial ureter identification (minutes) | 1 day (day of surgery)
  Measurement of the average time required for initial ureter identification (minutes)
Fraction of cases for which ureter integrity status (leak vs. no leak) and function (flow/obstructions) were determined at closing without the need for invasive procedures and/or tissue manipulation | 1 day (day of surgery)
  Measure the proportion of cases for which ureter integrity status (leak vs. no leak) and function (flow/obstructions) were determined at closing without the need for invasive procedures and/or tissue manipulation
Among cases that normally require ureter skeletonization/ureter dissection, the proportion of cases where skeletonization/ureter dissection could be reduced or eliminated | 1 day (day of surgery)
  Measure the fraction of cases where skeletonization/ureter dissection could be reduced or eliminated in cases where ureter skeletonization/ureter dissection are normally required
Average time period of ureter visualization provided by the first dose of Nizaracianine | 1 day (day of surgery)
  Measure the average time period of ureter visualization provided by the first dose of Nizaracianine
Average dose interval and average number of doses of Nizaracianine preferred by surgeons for optimal visualization of the ureters during surgeries of various lengths (Phase 3 only) | 1 day (day of surgery)
  Measure the average dose interval and average number of doses of Nizaracianine preferred by surgeons for optimal visualization of the ureters during surgeries of various lengths (Phase 3 only)
Among subjects with ureter injury, the proportion of cases detected intraoperatively | 1 day (day of surgery)
  Among subjects with ureter injury, measure the fraction of cases detected intraoperatively
Among subjects with intraoperative detection of ureter injury, the proportion of cases in which Nizaracianine assisted repair | 1 day (day of surgery)
  Among subjects with intraoperative detection of ureter injury, measure the fraction of cases in which Nizaracianine assisted repair
For a particular surgical procedure type, average overall surgery time (Phase 3A only) | 1 day (day of surgery)
  Measure the average overall surgery time for a particular surgical procedure type (Phase 3A only)

OTHER OUTCOMES:
In Phase 3A, comparison of the primary outcome measure between treatment and control arms | 1 day (day of surgery)
  In Phase 3A, compare the proportion of subjects for whom the surgeon is able to successfully identify the required length of the ureters (specified prior to surgery by the surgeon) with a peak signal-to-background ratio (SBR) ≥ 1.5 between the treatment and control arms.
In Phase 3B, comparison of the primary outcome measure between NIR imaging and white light imaging in the same subject | 1 day (day of surgery)
  In Phase 3B, compare the proportion of subjects for whom the surgeon is able to successfully identify the required length of the ureters (specified prior to surgery by the surgeon) with a peak signal-to-background ratio (SBR) ≥ 1.5 for NIR imaging versus white light imaging in the same subject
In bladder-involved cases, the fraction of cases where Nizaracianine helped identify bladder anatomy | 1 day (day of surgery)
  Calculation of the fraction of cases where Nizaracianine helped identify bladder anatomy in bladder-involved surgery cases
The proportion of cases where Nizaracianine provided NIR fluorescence enhancement of blood vessels in the surgical field | 1 day (day of surgery)
  Measurement of the fraction of cases where Nizaracianine provided NIR fluorescence enhancement of blood vessels in the surgical field

CONTACTS AND LOCATIONS:
Overall Officials: John V Frangioni, M.D., Ph.D., Study Chair — Curadel Surgical Innovations, Inc. (CSI); John V Frangioni, M.D., Ph.D., Study Director — Curadel Surgical Innovations, Inc. (CSI); Alexander L Vahrmeijer, M.D., Ph.D, Principal Investigator — Leiden University Medical Centre (LUMC)
Locations (8):
- United States (3):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Board of Trustees of Leland Stanford Junior University, Redwood City, California
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
- Netherlands (5):
  - University Medical Center Groningen, Groningen
  - Martini Hospital, Groningen
  - Leiden University Medical Centre (LUMC), Leiden
  - Erasmus Medical Centre, Rotterdam
  - Isala Zwolle, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Valk KS, Handgraaf HJ, Deken MM, Sibinga Mulder BG, Valentijn AR, Terwisscha van Scheltinga AG, Kuil J, van Esdonk MJ, Vuijk J, Bevers RF, Peeters KC, Holman FA, Frangioni JV, Burggraaf J, Vahrmeijer AL. A zwitterionic near-infrared fluorophore for real-time ureter identification during laparoscopic abdominopelvic surgery. Nat Commun. 2019 Jul 16;10(1):3118. doi: 10.1038/s41467-019-11014-1. PMID 31311922